CLINICAL TRIAL: NCT01744847
Title: DGT Versus TPS in Patients With Initial PD Cannulation by Chance; Prospective Randomized Multi-center Study
Brief Title: DGT Versus TPS in Patients With Initial PD Cannulation by Chance; Prospective Multi-center Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Soon Chun Hyang University (Other)
Responsible Party: Principal Investigator, Lee Woong Cheul, fellow of gastroenterology, Soon Chun Hyang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD-2012-010
Record Dates: First submitted 2012-11-09; First posted 2012-12-07 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Pancreatitis; Cholangitis; Cholecystitis
MeSH Terms: conditions — Pancreatitis; Cholangitis; Cholecystitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DGT, Tracer Metro® Direct™ Wire Guide (Active Comparator): Double guide wire technique was performed by Tracer Hybrid® Wire Guides and Tracer Metro® Direct™ Wire Guide
  Interventions: Device: Tracer Hybrid® Wire Guides, Tracer Metro® Direct™ Wire Guide
- TPS, Tracer Hybrid® Wire Guides (Active Comparator): trans pancreatic sphincterotomy was performed by Tracer Hybrid® Wire Guides
  Interventions: Device: Tracer Hybrid® Wire Guides, Tracer Metro® Direct™ Wire Guide

INTERVENTIONS:
Device: Tracer Hybrid® Wire Guides, Tracer Metro® Direct™ Wire Guide — one guide wire insert to the pancreatic duct and other guide wire insert to the Common bilde duct for cannulation
  Other Names: Tracer Hybrid® Wire Guides; Tracer Metro® Direct™ Wire Guide

SUMMARY:
In patients with pancreatic duct cannulation initially by chance, double guide wire technique and trans pancreatic sphincterotomy facilitate biliary cannulation and show the similar success rates. The incidence of post-procedure pancreatitis was similar in the two groups, but post-procedure hyperamylasemia was significantly higher in the DGT group.

DETAILED DESCRIPTION:
This was a prospective, randomized study conducted in three tertiary referral hospital in Korea. Three endoscopists performed the ERCP who had ERCP experience more than ten years From October 2010 to August 2012, ERCPs were performed on patients with pancreatobiliary diseases at Soonchunhyang University Seoul Hospital, Hanyang University Guri Hospital and Kosin University Gospel Hospital. Bile duct cannulation was attempted for various reasons (removal of bile duct stones, biliary stenting, cytology of bile, biopsy of the bile duct, etc.).

Patients who satisfied the following inclusion criteria were enrolled in this study: (1) initially pancreatic duct cannulation by chance, (2) successful insertion of the guidewire into the pancreatic duct to at least half of the presumed total length of the pancreatic duct,, and (3) age 20 years or older. Exclusion criteria were: (1) refusal the ERCP, (2) previous endoscopic sphincterotomy or endoscopic papillary balloon dilatation, (3) acute pancreatitis at the time of the procedure, (4) pregnancy and (5) anatomical change due to past surgery; total gastrectomy, Billroth II operation, Whipples's operation etc. Patients who satisfied the inclusion criteria were randomly assigned to either the double-guidewire technique (DGT) group or the transpancreatic precut sphincterotomy (TPS) group; A randomization list for group allocation was generated by using computer-based pseudo-random number generators. We compared both techniques , for a maximum of ten extra attempts which are CBD cannulation by each methods. We obtained the written informed consent from all enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

* ERCP patient, over 20 years old, pancreatic duct cannulation patients by chance

Exclusion Criteria:

* refuse the ERCP, post procedure state(EST, subtotal gastrectomy, Whipples' Op except gastroduodenostomy), use another method, under 20 years old.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2005-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
success rate between DGT and TPS | up to 22months
  from October 2010 to August 2012

SECONDARY OUTCOMES:
median cannulation time between DGT and TPS | during precedure time
  median time for precedure

OTHER OUTCOMES:
pancreatitis rate between DGT and TPS | upto 1 week
  We observation for the comlication upto 1 week after ERCP

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Digestive Research, Digestive Disease Center, Department of Internal Medicine, Soonchunhyang University College of Medicine, Soonchunhyang University Hospital, Seoul, Yongsan-gu, South Korea